CLINICAL TRIAL: NCT04256161
Title: Measurements of Sexual Steroids' Concentrations in Prostatic Tissue From Samples Taken by Biopsy Needle on Fresh Operating Parts : Measurements' Reliability
Brief Title: Measurements of Sexual Steroids' Concentrations in Prostatic Tissue
Acronym: Pré-HORM
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_0049
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
Keywords: Steroids' concentrations; Biopsy needle; Cystoprostatectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 sample of prostate tissue obtained by punch (90 mg) 6 samples of prostate tissue obtained by biopsy needle (3 mg by sample)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the investigators's previous work, measurements of intra-prostatic concentrations of sex steroids were determined on samples taken from the operating room using a punch.

In order to study the in-vivo intra-prostatic concentrations of sex steroid, it is necessary to validate a measurement technique performed on samples obtained by a biopsy needle used in standard care for prostate biopsy punctures allowing the diagnosis and follow-up of prostate cancer.

The aim of this project is to validate this measurement technique carried out on samples obtained by the biopsy needle and to define the optimal number of carrots obtained by biopsy offering dosage results comparable to the punch.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* With a bladder cancer
* Should be operated by total cystoprostatectomy at Foch Hospital
* Affiliated to a health insurance scheme
* Having expressed the non-opposition for the participation to the study

Exclusion Criteria:

* Patient receiving or has received a treatment by analog or antagonist of Luteinizing Hormone Releasing Hormone (LHRH), antiandrogens (steroidal or non-steroidal), 5 alpha-reductase inhibitor, docetaxel or cabazitaxel chemotherapy, abiraterone acetate, enzalutamide or corticosteroids
* Patient who does not understand French
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male with a bladder cancer and expected to benefit from a total cystoctoectomy in the Urology Department of Foch Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Intra-prostatic concentrations of sex steroids | Day 0
  To compare intra-prostatic concentrations of sex steroids on samples taken by punch (reference technique) and by an increasing number (1 to 3 carrots) of samples taken by biopsy needle (experimental technique) on fresh surgical specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Yann NEUZILLET, PhD, Principal Investigator — Hopital Foch, Suresnes
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No